CLINICAL TRIAL: NCT05436197
Title: The Expansion of a Parent-focused Physical Literacy Intervention for Early Childhood Called PLAYshop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Victoria (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLAYshop Expansion
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Motor Activity; Parent-Child Relations; Child Development
Keywords: Questionnaires; Semi-structured Interviews
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will complete the baseline measure and then be randomly assigned to group 1 (intervention) or group 2 (control), in a computer generated 1:1 sequence.
Masking Description: Participants: While the families will not be told explicitly if they have been assigned to the intervention or control group, they may be able to determine their group based on when their workshop is scheduled (i.e., immediately versus after completion of all study measures).
  Research Coordinator: The research coordinator will be aware of the group allocations as they will be in charge of coordinating random assignment and have to schedule participants into workshops and other measures based on their specific allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLAYshop Intervention (Experimental): Participants will receive a 60 minute virtual/hybrid physical literacy workshop, an equipment goody-bag with basic play equipment and printed resources, and access to a digital app with an online toolkit and four bi-weekly boosters lessons.
  Interventions: Behavioral: PLAYshop Program
- Control (No Intervention): Participants will receive the 60 minute virtual/hybrid physical literacy workshop, equipment goody-bag, and access to the digital app after completing the follow-up measures.

INTERVENTIONS:
Behavioral: PLAYshop Program — The intervention includes: 1. Educational Training - the 60 min virtual/hybrid workshop will be delivered by a trained facilitator. Parents will be introduced to physical literacy via education, group discussion, and active participation in fundamental movement skills (FMS) based activities with their child. 2. Distribution of Education Resources- Parents will be provided with physical literacy and physical activity printed resources. 3. Material resources -parents will also be provided a bag of inexpensive active play equipment (e.g., ball, bean bag, balloons). 4. Provide Follow-up Support- After the workshop, participants will gain access to an app with an online toolkit including new active play ideas, tips, and equipment they can make at home for active play. Additionally, participants will receive four bi-weekly booster lessons that include key workshop messages, support and encouragement for parents, reflection and check-in questions, and new activities to try with their child.
  Arms: PLAYshop Intervention

SUMMARY:
The PLAYshop program is a novel, brief, theory-based, parent-focused physical literacy intervention, that can help mitigate the impacts of the COVID-19 pandemic on physical activity of children from diverse and vulnerable families who have been disproportionally affected by the COVID-19 Pandemic.

Primary Research Question: Among vulnerable families (e.g., lower socioeconomic status), does the PLAYshop program increase parental capability, opportunity, and motivation to support preschool-aged children's physical literacy development, compared to controls?

DETAILED DESCRIPTION:
The overall objective of this study is to generate evidence for the efficacy of the PLAYshop program in diverse and vulnerable populations, such as families of lower socioeconomic status, who have been disproportionally affected by the COVID-19 Pandemic.

Research Questions:

Primary: Among vulnerable families (e.g., lower socioeconomic status), does the PLAYshop program increase parental capability, opportunity, and motivation to support preschool-aged children's physical literacy development, compared to controls? Secondary: What is the level of, and factors that influence, implementation at the family and program delivery level when working with vulnerable families? Tertiary: Does the PLAYshop program increase preschool-aged children's motivation and enjoyment, compared to controls?

Hypothesis for the primary research question: Increases in parental outcomes, including capability, opportunity, and motivation, will be greater in the intervention group, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children aged 3 to 5 years who live in the provinces of Alberta and British Columbia and meet at least one of the following criteria:

   * Statistics Canada's low income before tax cut-off based on household size and the population of the municipality they live in
   * have an education level below a bachelor's degree (participating parent)
   * are unemployed (participating parent)
   * are a single adult in their household
   * are connected with an agency partner that supports vulnerable populations
2. Research staff and any organization partners who lead the workshop

Exclusion Criteria:

1) Parents:

* who do not have internet access to complete the questionnaires and join the virtual workshop. This includes access to a device such as a smartphone, tablet, or laptop/computer and a data plan or WIFI.
* who are not comfortable reading, writing, speaking and listening to at least one the following languages: English, Spanish, Farsi, Mandarin (Simplified Chinese), or Cantonese (Traditional Chinese).
* that have participated in prior PLAYshop pilot and feasibility trials

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Change in parents' capability to support preschool-aged children's physical literacy development | Baseline (all), immediately after workshop (intervention), one week after baseline (control)
  Parental capability (i.e., knowledge), will be assessed via a parental questionnaire. This scale includes 9 items with values of 1-5; higher values mean more capability.
Change in parents' opportunity to support preschool-aged children's physical literacy development | Baseline (all), immediately after workshop (intervention), one week after baseline (control)
  Parental opportunity (e.g., perceived availability of resources (1 item), perceived barriers (5 items)) will be assessed via a parental questionnaire. Items have values of 1-5; higher values mean less parental opportunity. Citation for perceived barriers: Heitzler et al., 2006
Change in parents' motivation to support preschool-aged children's physical literacy development | Baseline (all), immediately after workshop (intervention), one week after baseline (control)
  Parental motivation (i.e., confidence (11 items), beliefs (4 items), outcome expectations (3 items), intentions (2 items), perceived behavioural control (4 items)) will be assessed via a parental questionnaire. Citation for beliefs and outcome expectations: Heitzler et al., 2006. Items have values of 1-5; higher values mean more parental motivation.

SECONDARY OUTCOMES:
Implementation: satisfaction and perceived usefulness (questionnaire) | Intervention group: Immediately after the workshop
  Satisfaction and perceived usefulness of the intervention will be assessed via a parental questionnaire in the intervention group only. This scale includes 3 items with values of 1-5; higher values mean more satisfaction and perceived usefulness.
Implementation: satisfaction and perceived usefulness (parental interview) | Intervention group: 2-month follow-up
  Satisfaction and perceived usefulness of the intervention will also be explored via brief semi-structured interviews with parents from the intervention group.
Implementation: facilitators and barriers (parental interview) | Intervention group: 2-month follow-up
  Implementation facilitators and barriers will be explored via brief semi-structured interviews with parents from the intervention group.
Implementation: facilitators and barriers (workshop leader interview) | At study completion, approximately 1 year from first workshop.
  Implementation facilitators and barriers will be explored via brief semi-structured interviews with workshop leaders.
Implementation: dose (parental interview) | Intervention group: 2-month follow-up
  The dose of the intervention will be explored via brief semi-structured interviews with parents from the intervention group.
Implementation: dose (app check-in questions) | Intervention group: Bi-weekly after workshop (i.e., 1, 3, 5, and 7 weeks)
  The dose of the intervention will be assessed via check-in questions as part of the booster lessons in the intervention group.
Implementation: dose (app usage data) | Intervention group: 2-month follow-up
  The dose of the intervention will be assessed via tracking of app usage in the intervention group.

OTHER OUTCOMES:
Change in children's motivation and enjoyment | Baseline (all), immediately after workshop (intervention), one week after baseline (control)
  Children's motivation and enjoyment will be assessed via a parental questionnaire that includes items from the Preschool Physical Literacy Assessment (Pre PLAy). This scale includes 4 items with values of 1-5; higher values mean more motivation and enjoyment. Citation: Cairney et al. (2018)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Carson, PhD, Principal Investigator — University of Alberta; Patti-Jean Naylor, PhD, Principal Investigator — University of Victoria; Ryan Rhodes, PhD, Principal Investigator — University of Victoria; Sam Liu, PhD, Principal Investigator — University of Victoria
Locations (1):
- Faculty of Kinesiology, Sport, and Recreation, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
To protect participant's personal data, IPD will not be shared with researchers outside of the research team.

REFERENCES:
- [Background] Heitzler CD, Martin SL, Duke J, Huhman M. Correlates of physical activity in a national sample of children aged 9-13 years. Prev Med. 2006 Apr;42(4):254-60. doi: 10.1016/j.ypmed.2006.01.010. Epub 2006 Feb 20. PMID 16490241
- [Background] Cairney J, Clark HJ, James ME, Mitchell D, Dudley DA, Kriellaars D. The Preschool Physical Literacy Assessment Tool: Testing a New Physical Literacy Tool for the Early Years. Front Pediatr. 2018 Jun 7;6:138. doi: 10.3389/fped.2018.00138. eCollection 2018. PMID 29930933